CLINICAL TRIAL: NCT03944681
Title: Gender Influence on Torsadogenic Actions of Droperidol Used as Postoperative Nausea and Vomiting Prophylaxis.
Brief Title: Gender Influence on Torsadogenic Actions of Droperidol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Clinical Professor, Head of Department of Anaesthesiology and Intensive Care, Medical University of Gdansk
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KB01
Record Dates: First submitted 2019-01-30; First posted 2019-05-09 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Arrhythmia, Droperidol
Keywords: postoperative nausea and vomiting; torsadogenic action; transmural dispersion of repolarisation; corrected QT interval
MeSH Terms: conditions — Arrhythmias, Cardiac; Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Droperidol group (Other): Droperidol (Xomolix, Kyowa Kirin) 1.25 mg i.v. bolus
  Interventions: Drug: Droperidol Injectable Solution

INTERVENTIONS:
Drug: Droperidol Injectable Solution — An electrocardiogram analysis in: 5,10,15,20 minutes after injection of 1.25 mg of droperidol used as PONV prophylaxis.
  Other Names: electrocardiogram analysis

SUMMARY:
Postoperative nausea and vomiting (PONV) is a quite common complication affecting patients undergoing general anesthesia. There are a few pharmacological agents of well known effectiveness in reducing the risk of PONV. One of them is droperidol, which is a butyrophenone derivant. It has been widely used for the prevention and treatment of PONV due to its high effectiveness and low cost. Though, droperidol has a relevant side effect, that is a repolarization prolongation. This can lead to life-threatening cardiac arrhythmias: polymorphic ventricular tachycardia (torsades de pointes, TdP) that can degenerate into ventricular fibrillation and cardiac arrest. This was a reason why in 2001 the FDA issued a "black box" warning on droperidol. Ever since papers focused on this problem have described the influence of small doses of droperidol on TdP genesis as weak. This could be explained by the fact, that QT/QTc (corrected QT) interval prolongation, which represents prolonged cardiac repolarization on ECG, is not the sole determinant of a drug's potential to cause arrhythmia. Another electrocardiographical marker of torsadogenic action is increased transmural dispersion of repolarization (TDR). TDR represents differences in the repolarization between myocardial "layers" (like epicardium, endocardium, myocardium cells). It is believed that the induction of QT/QTc lengthening must coexist with TDR increase at the same time to promote torsadogenic changes.

It has been known, on the basis of research, that females have been more potent to torsadogenic actions of pharmacological agents than males. That could be related to estrogen influence on ECG parameters, which had been proven on animal model. It hasn't been investigated, whether gender is an important factor when considering droperidol's torsadogenic potential.

The aim of this study is to answer a hypothesis, that women are more potent to torsadogenic actions of droperidol in comparison with men.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years old
* ASA (American Society of Anaesthesiologists) physical status 1 and 2

Exclusion Criteria:

* lack of informed consent
* ASA (American Society of Anaesthesiologists) physical status 3 and more
* admittance of repolarisation affecting drugs like: antiarrhythmics (Williams group I-IV), psychotropics, macrolides, antireflux drugs
* ischaemic heart disease
* cardiac failure NYHA (Hew York Heart Association) 1 and more
* congenital or acquired heart defects
* arrhythmias in anamnesis
* hormonal contraception,
* postmenopausal
* neoplasms

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
QT and corrected QT interval time | Change from baseline QT and corrected QT interval time at 5,10,15 and 20 minutes after administration of 1.25 mg droperidol
  measured in milliseconds
Time interval between T wave peak and T wave end | Change from baseline T peak - T end time at 5,10,15 and 20 minutes after administration of 1.25 mg droperidol.
  measured in milliseconds

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Owczuk, Professor, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No